CLINICAL TRIAL: NCT06799338
Title: Real World Use of Lenacapavir, as an add-on to an Optimized Background Regimen in France: a Retrospective Observational Study (LENAddOn)
Brief Title: Real World Use of Lenacapavir, as an add-on to an Optimized Background Regimen in France
Acronym: LENAddON
Status: Recruiting | Type: Observational
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Other Study IDs: CREPATS 20
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: HIV I Infection
MeSH Terms: interventions — lenacapavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LENAddOn is a retrospective, observational, national, multicenter study: Data will be collected from medical records in 21 centers, and captured with a dedicated eCRF created on the study purpose.
  Patients will be included if they initiated LEN from 20 June 2023 to 30 June 2024.
  All collected data are routinely reported by clinicians in medical records. All clinical decisions All collected data are routinely reported by clinicians in medical records, and will be collected using a dedicated electronic case report form (eCRF) created on this purpose, to ensure confidentiality of data.
  Interventions: Drug: Lenacapavir Injection

INTERVENTIONS:
Drug: Lenacapavir Injection — Patients will be included if they initiated LEN from 20 June 2023 to 30 June 2024.
  All collected data are routinely reported by clinicians in medical records. All clinical decisions All collected data are routinely reported by clinicians in medical records, and will be collected using a dedicated electronic case report form (eCRF) created on this purpose, to ensure confidentiality of data.

SUMMARY:
For most people with HIV (PWH), an effective antiretroviral regimen can be devised. However, some PWH have multiple treatment failures due to viral resistance or unacceptable side effects to medication and no longer have durable viral suppression. People with multidrug-resistant HIV-1 are at increased risk for hospitalization, progression to acquired immunodeficiency syndrome, and death.

Lenacapavir (LEN) is a first-in-class capsid inhibitor and has been evaluated through the CAPELLA phase 3 trial in PWH with replicative multidrug-resistant HIV-1. In this trial, LEN combined with an optimized background regimen (OBR) led to high levels of viral suppression, as more than 80% of participants achieved undetectable plasma HIV-RNA, associated with increasing in CD4 T cell counts.

LEN has become publicly available in France from June 20, 2023, and prescriptions are discussed and validated by multidisciplinary committees in the hospitals, including HIV physicians, virologists and pharmacologists.

From the time LEN was made publicly available in France, no real-world data have been generated to describe the real-world use of LEN, in association with an OBR, in various patient's profiles who may differ from the subjects included the CAPELLA trial.

Thus, investigators plan to conduct a national, multicenter, retrospective observational study to describe baseline socio-demographic, clinical and biological profiles of PWH receiving LEN + OBR in French real-world settings, to determine the continuation of LEN injections at weeks 26 and 52, and to determine the reasons for stopping LEN in case of no continuation of LEN injections.

In its current indication, LEN is reserved for a minority of PWH. However, France is the second-largest prescribing country for this drug, and one year after it was first marketed, it seems essential to review its use. Whether LEN injections are continued 6 and 12 months after starting treatment is a crucial question for understanding its use in treatment centers.

Lenacapavir has become publicly available in France in June 20, 2023. LEN prescriptions in France are discussed and validated by multidisciplinary committees, including HIV physicians, virologists and pharmacologists in the hospitals.

DETAILED DESCRIPTION:
For most people with human immunodeficiency virus type 1 (HIV-1) infection, an effective antiretroviral regimen can be devised. However, some PWH have multiple treatment failures due to viral resistance or unacceptable side effects to medication and no longer have durable viral suppression. People with multidrug-resistant HIV-1 are at increased risk for hospitalization, progression to acquired immunodeficiency syndrome, and death.

Lenacapavir (LEN) is a first-in-class inhibitor of HIV-1 capsid function.5 By interfering with capsid-mediated nuclear uptake of pre-integration complexes and impairing virion production, lenacapavir inhibits viral replication at both early and late stages of the life cycle. In vitro, lenacapavir has antiviral activity against viral mutations that are resistant to major antiretroviral classes of drugs. LEN can be administered in a long-acting fashion - up to every 6 months subcutaneously or weekly orally - because of its picomolar potency, low clearance, and slow release kinetics. Its efficacy has been demonstrated in the CAPELLA phase 3 trial. For the primary endpoint (following 14 days of functional monotherapy) of CAPELLA, 88% of participants randomized to LEN achieved a significant viral load reduction (≥0.5 log10 copies/mL decline) versus 17% on placebo (p< 0.001).10 Consistent with results through week 52 of the CAPELLA study, LEN combined with an optimized background regimen (OBR) continued to result in high and sustained rates of virologic suppression and increases in CD4 T cell counts through week. When analyzed as missing equals excluded, 82% of participants achieved HIV-1 RNA <50 copies/mL.

Lenacapavir has become publicly available in France in June 20, 2023. LEN prescriptions in France are discussed and validated by multidisciplinary committees, including HIV physicians, virologists and pharmacologists in the hospitals.

From the time LEN was made publicly available in France, no real-world data have been generated (except for a few clinical cases) to describe the real-world use of LEN, in association with an OBR, in various patient's profiles who may differ from the subjects included the CAPELLA trial.

To document the real-world use of LEN plus OBR, this study will describe baseline socio-demographic, clinical and biological profiles of PWH receiving LEN with OBR, and determine the continuation of LEN injections at week 26 and week 52 in real-life settings in France.

In its current indication, LEN is reserved for a minority of PWH. However, France is the second-largest prescribing country for this drug, and one year after it was first marketed, it seems essential to review its use. Whether LEN injections are continued 6 and 12 months after starting treatment is a crucial question for understanding its use in treatment centers.

LENAddOn is a retrospective, observational, national, multicenter study

This study consists in retrospectively analyzing data from participant medical records, without intervention. All clinical decisions are made as part of routine management, and are not protocolized. No additional clinical visits or biological samples are required for the study. For this reason, weeks 26 and 52 are for information only, but a window of +/- 2 weeks will be allowed for data capture. Initiation of LEN and optimization of associated ART is chosen by the physician, in agreement with the patient, after discussion within a multidisciplinary committee, as recommended by the guidelines. All these decisions are independent of the LENAddOn observational study.

All participants to be included in the study have already begun their LEN treatment, since the period for initiating LEN (first dose received) has ended (end of June 2024). They will be therefore identified retrospectively for inclusion in the study. Some patients will not have completed their 52-week follow-up at the time of inclusion in the study: their follow-up will be prospective. Nevertheless, data collection will be retrospective. Entry of participants' data into the eCRF will only be authorized for a period of time following the end of the follow-up period for the last patient included.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years);
* With HIV-1 infection;
* Who received a first dose of LEN (oral or injectable) with and OBR from the ending of the French national early access program (20 June 2023) to 30 June 2024;
* Who did not refuse the collection and use of their data.

Exclusion Criteria:

- HIV-2 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We anticipated about 120 patients initiating LEN from 20 June 2023 to 30 June 2024 in France.
  We plan to include 80 subjects, followed in 21 French centers.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure the number of participants who received lenecapavir injection | Week26
Measure the number of participants who received a lenacapavir injection | Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Romain PALICH, MD, Principal Investigator — Pitie-Salpetriere Hospital
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No